CLINICAL TRIAL: NCT01215526
Title: Effectiveness and Safety of Firmagon® in Androgen Ablative Therapy of Advanced Hormone-dependent Prostate Carcinoma in the Netherlands
Brief Title: A Study Into the Effectivity and Safety of Firmagon, Prescribed for Treatment of Patients With Advanced Prostate Cancer
Acronym: FAST-NL
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: FE200486 CS46
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients eligible for hormone ablation therapy who are prescribed Firmagon will be followed for a maximum of 3 years to estimate the progression free survival. Data on testosteron levels, QoL and LUTS will be collected if this information is available. Safety information (adverse events) will be collected.

ELIGIBILITY:
Inclusion Criteria:

- Patients with advanced hormone-dependent prostate carcinoma that are eligible for hormone therapy

Exclusion Criteria:

- Patients with a contraindication for prescription of Firmagon®

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2010-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To estimate the progression-free survival (PFS) failure rate | Maximum 3 years

SECONDARY OUTCOMES:
To enhance the knowledge on known undesirable effects under routine conditions and to obtain further knowledge about so far unknown and rare undesired effects | Every 3 months (during 3 years)
To prescribe the change in patient's quality of life (QoL) during therapy. | From study start and after 6 months
To assess the improvement of IPSS from baseline after 3 months of Firmagon therapy and at end-of-therapy | From study start, after 3 months and at end of treatment
To assess the reduction of prostate volume (neoadjuvant therapy) | Fom baseline after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (47):
- Netherlands (47):
  - Jeroen Bosch Ziekenhuis, locatie Carolus, 's-Hertogenbosch
  - Flevoziekenhuis, Almere Stad
  - Bovenij Ziekenhuis, Amsterdam
  - Wilhelminaziekenhuis, Assen
  - Rode Kruis Ziekenhuis, Beverwijk
  - Tergooiziekenhuizen, Blaricum
  - Amphia Ziekenhuis, Breda
  - Ljsselland Ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf Groep, Delft
  - Deventer Ziekenhuis, Deventer
  - Slingeland Ziekenhuis, Doetinchem
  - Alb.Schweitzer Ziekenhuis, loc. Dordwijk, Dordrecht
  - Gelderse Vallei, loc. Barneveld, Ede
  - Admiraal de Ruyter Ziekenhuis, Flushing
  - St. Anna Ziekenhuis, Geldrop
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Rivas Beatrixziekenhuis, Gorinchem
  - Het Groene Hart Ziekenhuis, Gouda
  - Buitenpolikliniek, Groenlo
  - Martini Ziekenhuis, Groningen
  - Ziekenhuis St Jansdal, Harderwijk
  - Elkerliek Ziekenhuis, Helmond
  - Tergooiziekenhuizen, Hilversum
  - Medisch Centrum Leeuwarden, Leeuwarden
  - LUMC, Leiden
  - Rijnland Ziekenhuis, Leiderdorp
  - MUMC, Maastricht
  - Ziekenhuis Bernhoven, loc. Oss, Oss
  - Waterland Ziekenhuis, Purmerend
  - Franciscus Ziekenhuis, Roosendaal
  - Havenziekenhuis, Rotterdam
  - Vlietland Ziekenhuis, Rotterdam
  - Orbis Medisch Centrum, Sittard-Geleen
  - Alb. Schweitzer Ziekenhuis loc. Sliedrecht, Sliedrecht
  - Antonius Ziekenhuis, Sneek
  - Ruwaard v Putten/vWeel Bethesda Zkhs, Spijkenisse
  - Zorgzaam Ziekenhuis, Terneuzen
  - Hagaziekenhuis loc. Leyweg, The Hague
  - Hagaziekenhuis loc. Sportlaan, The Hague
  - Ziekenhuis Rivierenland, Tiel
  - Antonius Ziekenhuis, loc. Oudenrijn, Utrecht
  - Diakonessenhuis Utrecht, Utrecht
  - Ziekenhuis Bernhoven, loc. Veghel, Veghel
  - Maxima Medisch Centrum, Veldhoven
  - St. Jans Gasthuis, Weert
  - Albert Schweitzer Ziekenhuis, Zwijndrecht
  - Isala Klinieken, Zwolle